CLINICAL TRIAL: NCT06435481
Title: Tolerability and Acceptance of Two Oral Hydrocortisone Compounding Formulation for Pediatrics
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HIDROGUM21; 2021-001069-20 (EudraCT Number)
Record Dates: First submitted 2024-04-29; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-04

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chewable Tablet Group (Experimental): Group of patients receiving a new hydrocortisone formulation in the form of chewable tablets. Patients in this group will take the 3D printed chewable tablets orally for a duration of three months.
  Interventions: Drug: 3D printed chewable formulation of hydrocortisone
- Oral Suspension Group (Active Comparator): Group of patients receiving the standard hydrocortisone formulation in the form of an oral solution. Patients in this group will orally ingest the solution over a period of three months.
  Interventions: Drug: Oral suspension of hydrocortisone

INTERVENTIONS:
Drug: 3D printed chewable formulation of hydrocortisone — Administration of a novel hydrocortisone formulation provided as chewable tablets. Each tablet, manufactured with a volume dosing device (3D printer), contains a precise dosage of hydrocortisone.
  Arms: Chewable Tablet Group
Drug: Oral suspension of hydrocortisone — Administration of a standard hydrocortisone oral suspension. The solution, based on simple syrup, contains 1mg of hydrocortisone per milliliter.
  Arms: Oral Suspension Group

SUMMARY:
The study aims to evaluate the tolerability and acceptance of two compounded formulations of hydrocortisone prepared in the Vall d'Hebron University Hospital (VHUH) Pharmacy Service: one, an oral suspension and the other, chewable tablets prepared using a volume dosing device (M3DIMAKER 3D printer). The main goal is to enhance patient care and adherence among pediatric patients.

This prospective, experimental study employs a randomized, crossover design and will take place solely at VHUH. Approximately 25-30 eligible patients diagnosed with adrenal hyperplasia, isolated primary adrenal insufficiency, or panhypopituitarism will be recruited. Each patient will receive each hydrocortisone formulation for a period of 3 months, totaling 6 months of treatment per patient. All patients will receive the medication at their usual dose and both formulations to assess tolerability and acceptance.

DETAILED DESCRIPTION:
Adrenal insufficiency arises from inadequate synthesis of adrenal hormones, with primary, secondary, or tertiary forms depending on the defect's location-adrenal, pituitary, or hypothalamic. Hydrocortisone (17-Hydroxycorticosterone) is the preferred cortisol replacement.

Pediatric hydrocortisone formulations are not commercially available in any presentation. Consequently, compounded formulations are prepared as standard practice. Vall d'Hebron University Hospital's Pharmacy Service currently provides a liquid hydrocortisone formulation for these patients. While liquid formulations are often preferred due to their better dose adjustment and improved acceptability by pediatric patients, they have limitations such as shorter shelf life, possible special storage conditions, and taste problems due to bitter active ingredients. In some cases, particularly for chronic treatments with established and constant doses, other options such as capsules may be considered. Capsules offer longer stability, longer expiration dates, and do not require special storage conditions.

In this context, this study aims to determine the tolerability and acceptance of a new solid magistral formula in the form of chewable hydrocortisone tablets, prepared using a volume dosing device (M3DIMAKERTM 3D printer), compared to the usually preferred liquid formulation. Each of the formulations will be administered for three months. Evaluating the results will allow us to improve assistance to pediatric patients by offering the formulation with better tolerability and acceptance. The study will take place at Vall d'Hebron University Hospital, led by the Pharmacy Service in collaboration with the Pediatric Endocrinology Service.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of both sexes, ≥ 6 years old without swallowing problems and up to 17 years old, at the time of signing the informed consent document by parent(s) or guardian(s) and/or patients.
* Diagnosis of adrenal hyperplasia or isolated primary adrenal insufficiency or panhypopituitarism (secondary or tertiary adrenal insufficiency).

Exclusion Criteria:

* Known hypersensitivity to any of the excipients in the formulation of hydrocortisone.
* Any disorder or situation (decompensation) that, in the opinion of the investigating physician, poses a risk of non-compliance with the treatment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Tolerability and acceptance of the two compounded oral hydrocortisone formulations | 6 months
  Tolerability will be assessed using a five-point questionnaire, while acceptability will be measured using the hedonic facial scale.

SECONDARY OUTCOMES:
Efficacy, compliance and safety of each hydrocortisone formulation | 6 months
  Efficacy will be assessed by the variation in hydrocortisone dosage as a percentage compared to the previous visit, the presence of intercurrent issues, and emergency room visits resulting from the underlying condition.
  Treatment adherence will be estimated through monitoring medication dispensations from the Pharmacy Service and counting returned medication.
  Safety will be evaluated by reporting potential adverse effects of treatment, the presence of intercurrent issues, and emergency room visits during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hospital Universitari Vall d'Hebron, Study Chair — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No